CLINICAL TRIAL: NCT03964948
Title: Development of Novel MRI Methods for Detecting and Measuring Renal Injury/Fibrosis
Brief Title: Kidney Fibrosis and MRI
Acronym: ARCF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-4428
Record Dates: First submitted 2019-05-20; First posted 2019-05-28 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy Volunteers (Other): 20 healthy volunteers will be recruited and will receive a kidney MRI and the same blood and urine labs that are collected for the other arms. Results will be compared to the disease groups.
  Interventions: Diagnostic Test: Kidney MRI
- Kidney Transplant (Other): 20 subjects that have received a kidney transplant that have had a biopsy performed within the past 12 months will be enrolled. They will receive a kidney MRI and will have blood and urine collected.
  Interventions: Diagnostic Test: Kidney MRI
- Stage 2-5 CKD (Other): 20 subjects that have been diagnosed with stage 2-5 CKD and have had a biopsy performed within the past 12 months will be enrolled. They will receive a kidney MRI and will have blood and urine collected.
  Interventions: Diagnostic Test: Kidney MRI
- Lupus nephritis (Other): 20 subjects that have that have active lupus nephritis and have had a biopsy performed within the past 12 months will be enrolled. They will receive a kidney MRI and will have blood and urine collected.
  Subjects that are post-lupus treatment will receive an additional MRI at the time of the next biopsy.
  Interventions: Diagnostic Test: Kidney MRI

INTERVENTIONS:
Diagnostic Test: Kidney MRI — An MRI examination will be completed per research MRI protocol.

SUMMARY:
The investigators plan a prospective cross-sectional study of pediatric and adult healthy volunteers and patients with chronic kidney disease that will correlate a variety of quantitative MRI biomarkers with severity of renal insufficiency and available histopathology. Over 3 years, the investigators will recruit approximately 20 healthy volunteers, 20 patients with chronic kidney disease (CKD) Stage 2-5, and 20 patients with renal transplant kidneys. The investigators also plan to assess the effect of inflammation on the quantitative MRI biomarkers by recruiting approximately 20 additional patients with active lupus nephritis.

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all of the following criteria will be eligible for the study:

1. ≥ 10 and ≤ 25 years of age and;
2. Kidney transplant patients, who have had a recent kidney biopsy (within 1 year) that shows interstitial fibrosis OR
3. Patients with CKD Stage 2-5 who have previously had a biopsy (within 1 year) OR
4. Lupus patients with active nephritis who will undergo biopsy evaluation before and after induction therapy OR
5. Healthy Controls

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Known contraindication to MR imaging (e.g., implanted non-MRI compatible device)
2. Known or suspected pregnancy. Female subjects of child bearing potential will undergo a urine pregnancy test prior to imaging.
3. Inability to undergo MRI without sedation/anesthesia.
4. Non-English Speaking

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Development of noninvasive MRI methods to measure kidney disease using MR elastography. | 3 years
Development of noninvasive MRI methods to measure kidney disease using quantitative T1 mapping. | 3 years
Development of noninvasive MRI methods to measure kidney disease using T1rho mapping. | 3 years
Development of noninvasive MRI methods to measure kidney disease using T2 mapping. | 3 years
Development of noninvasive MRI methods to measure kidney disease using magnetization transfer imaging. | 3 years
Development of noninvasive MRI methods to measure kidney disease using diffusion-weighted imaging. | 3 years
  Intra-voxel incoherent motion and diffusion tensor imagining will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided